CLINICAL TRIAL: NCT01486433
Title: An Open-Label, Randomized, 2-Way Crossover Study to Evaluate the Effect of Multiple Doses of Epanova® on the Multiple-Dose Pharmacokinetics of Simvastatin in Healthy Normal Subjects
Brief Title: The Effect of Multiple Doses of Epanova® on the Multiple-Dose Pharmacokinetics of Simvastatin in Healthy Normal Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OM-EPA-007
Record Dates: First submitted 2011-11-29; First posted 2011-12-06 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Hypertriglyceridemia
Keywords: eicosapentaenoic acid; docosapentaenoic acid; arachidonic acid; hypertriglyceridemia; simvastatin
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Simvastatin; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epanova and Simvastatin (Experimental)
  Interventions: Drug: Simvastatin; Drug: acetylsalicylic acid (ASA); Drug: omefas
- Simvastatin (Active Comparator)
  Interventions: Drug: Simvastatin; Drug: acetylsalicylic acid (ASA)

INTERVENTIONS:
Drug: Simvastatin — 40 mg (1 tablet) simvastatin once a day
Drug: acetylsalicylic acid (ASA) — 81 mg aspirin (1 tablet), once a day, co-administered with simvastatin
  Other Names: aspirin
Drug: omefas — 4 g (4 capsules) Epanova once a day, co-administered with simvastatin and aspirin
  Other Names: Epanova
  Arms: Epanova and Simvastatin

SUMMARY:
The primary objective is to determine the effect of multiple doses of Epanova® (omega fatty acids) on the pharmacokinetics (PK) of multiple 40 mg doses of simvastatin.

DETAILED DESCRIPTION:
The study is testing the hypothesis that there is no interaction between Epanova and concomitant administration of simvastatin and aspirin. No drug interaction will be claimed if, following concomitant administration of simvastatin, aspirin and Epanova or only simvastatin and aspirin, the 90% confidence intervals (CIs) for the geometric mean ratios (GMRs) of the back-transformed PK parameters, area under the plasma concentration versus time curve (AUC0-tau) and concentration at the end of a dosing interval (Cmax,ss), for simvastatin and beta- hydroxysimvastatin acid,fall within 80%-125%.

ELIGIBILITY:
Inclusion Criteria:

Subjects must fulfil all of the following inclusion criteria to be eligible for participation in the study, unless otherwise specified:

1. Healthy adult male or female volunteers, 18-55 years of age, inclusive.
2. Body mass index (BMI) ≥ 18 and ≤ 29.9 (kg/m2).
3. Medically healthy with clinically insignificant screening results. Hemoglobin must be ≥ the lower limit of normal.
4. Continuous non-smokers who haven't used nicotine-containing products for at least 6 months prior to the first dose.
5. Voluntarily consent to participate in the study and to follow the restrictions and procedures outlined for the study.
6. Females must be of non-childbearing potential, and have undergone sterilization procedures at least 6 months prior to the first dose or be postmenopausal with amenorrhea for at least 2 years prior to first dosing and follicle stimulating hormone (FSH) serum levels ≥ 40 mIU/mL.

Exclusion Criteria:

Subjects may be excluded from the study if there is evidence of any of the following criteria at screening, check-in, or at any time during the study, as appropriate:

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, haematological, gastrointestinal (GI), endocrine, immunologic, dermatologic, neurological, or psychiatric disease in the opinion of the PI.
2. Personal or familial history of bleeding disorder(s), thromboembolic disease, clinical GI bleeding, or any history of GI surgery except uncomplicated appendectomy or cholecystectomy, or colorectal surgery for polyps, nonmalignant tumors, or diverticula.
3. Positive urine drug/alcohol testing at screening or check-in.
4. Positive result for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV).
5. History or presence of alcoholism or drug abuse within the past 2 years.
6. Subject has been on a special diet (for whatever reason) within the 28 days prior to the assigned first dose of study drug or anytime during the study.
7. Known sensitivity or allergy to soybeans, fish, and/or shellfish.
8. Hypersensitivity or idiosyncratic reaction to compounds related to simvastatin (i.e., HMG-CoA reductase inhibitors) and/or Epanova® and/or aspirin.
9. Subject is a female who is pregnant or lactating.
10. Use of any prescription medication within 14 days prior to the first dose.
11. Use of any over-the-counter (OTC) medication, including herbal products (e.g., bromelains, danshen, dong quai [Angelica sinensis], garlic, ginko biloba, ginseng, and St. John's wort, NSAIDs), vitamin K or food supplements (especially omega-3-fatty acids) within the 7 days prior to first dosing.
12. Use of any drugs known to significantly inhibit [strong or moderate] or induce liver enzymes involved in drug metabolism [CYP P450]) within 30 days prior to check-in.
13. Donation of blood or significant blood loss within 56 days prior to check- in.
14. Donation of plasma within 7 days prior to check-in.
15. Participation in another clinical trial within 30 days prior to check-in.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2011-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC0-tau) | 14 days
  Area under the plasma concentration versus time curve (AUC0-tau)for simvastatin and beta- hydroxysimvastatin acid, measured over the 24 hour period after the 14th dose
Concentration at the end of a dosing interval (Cmax,ss) for simvastatin and beta- hydroxysimvastatin acid, | 14 days
  Maximum measured plasma concentration for simvastatin and beta- hydroxysimvastatin acid,during the 0-24 hour dosing interval for the 14th simvastatin dose (Day 14)measured over the 24 hour period after the 14th dose.

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Davidson, MD, FACC, Study Director — Omthera Pharmaceuticals, Inc
Locations (1):
- Tempe, Arizona, United States